CLINICAL TRIAL: NCT05446584
Title: Pathways Relating Amnestic MCI to a Mild Traumatic Brain Injury History
Acronym: PATH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christian Lobue, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: STU-2022-0591
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment; Amnestic Mild Cognitive Disorder; Amnestic Mild Cognitive Impairment; Mild Traumatic Brain Injury; Concussion, Brain
Keywords: MCI; TBI; memory; biomarker; Alzheimer
MeSH Terms: conditions — Cognitive Dysfunction; Brain Concussion

STUDY DESIGN:
Intervention Model Description: All subjects will complete 3 conditions of HD-tDCS. Each HD-tDCS condition is comprised of 3 days of active or sham stimulation targeting the left frontal and temporal lobes (i.e., within-subjects design), randomized by order, and separated by 14 days to avoid carry-over effects.
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be informed that sham and active HD-tDCS will be used in the study, but they will be masked to condition. Aside from the PI, other study team members who perform assessments will be masked to HD-tDCS condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active left frontal HD-tDCS (Active Comparator): Electrodes will be placed in a 4x1 ring configuration over the frontal region in accordance with the International 10-10 EEG system. Stimulation will consist of a ramp up period in which the electrical current is gradually increased, 30 minutes of stimulation at 2 mA, and a ramp down period during which the electrical current is gradually removed. Stimulation will be applied back-to-back over three consecutive days.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation
- Active left temporal HD-tDCS (Active Comparator): Electrodes will be placed in a 4x1 ring configuration over the left temporal region in accordance with the International 10-10 EEG system. Stimulation will consist of a ramp up period in which the electrical current is gradually increased, 30 minutes of stimulation at 2 mA, and a ramp down period during which the electrical current is gradually removed. Stimulation will be applied back-to-back over three consecutive days.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation
- Sham HD=tDCS (Sham Comparator): Electrodes will be placed in the same 4x1 ring configuration over the frontal region as the active left frontal condition to ensure a useful control condition. Stimulation will consist of a 30-second ramp up period until reaching 2 mA, followed immediately by a 30-second ramp down, and off for 29 minutes. The same ramp up and down process will be repeated in the final minute of the session to help preserve masking of conditions. Sham stimulation will be applied back-to-back over three consecutive days.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High Definition Transcranial Direct Current Stimulation — HD-tDCS for this study is not intended to be a treatment, and will be applied continuously for 30 minutes at sham (0 mA) or 2 mA for active conditions across 3 consecutive daily sessions to probe neural circuit integrity. This specific HD-tDCS device is completely computer driven, running on a laptop using specialized software. Circular electrodes (12-mm in diameter) filled with conductive gel will be placed in a 4x1 ring configuration with the central electrode being the anode surrounded by four cathodes.

SUMMARY:
This study will probe if the biological changes in amnestic mild cognitive impairment (aMCI) are related to a history of mild traumatic brain injury (mTBI) using high definition transcranial direct current stimulation (HD-tDCS) and blood-derived biomarker tools. Participants who Do as well as those who Do Not have a history of mTBI will be enrolled in the study.

DETAILED DESCRIPTION:
Ten study visits will be completed by each participant. The initial visit will include a blood draw and a baseline memory evaluation. Afterwards, participants will be randomized to begin with one of 3 conditions of HD-tDCS. The three conditions are sham-control, active stimulation to frontal region, and active stimulation to left temporal region. All participants will be expected to completed each HD-tDCS condition, which will be counterbalanced and separated by 14 days. Active HD-tDCS will be applied at 2 mA for 30 minutes over 3 consecutive daily sessions while sham stimulation will be applied for the same duration and timespan. All subjects will complete memory assessments again immediately following each HD-tDCS condition for a total of four test sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Active diagnosis of amnestic mild cognitive impairment
2. Presence of an mTBI history for the mTBI+ group; absence of an mTBI history for a control sample
3. Female and male subjects
4. All races/ethnicities
5. Age 55 years and older
6. Fluent in English

Exclusion Criteria:

1. Mild traumatic brain injury within past year
2. Lifetime history of moderate or severe brain injury
3. Lifetime major neurologic syndromes (e.g., stroke, epilepsy, brain tumor)
4. Lifetime major cardiovascular conditions (e.g., heart attack, heart failure)
5. Current substance use disorder
6. Current major psychiatric disorders (e.g., major depressive disorder, bipolar disorder)
7. Current vision or hearing impairment that interferes with testing
8. Any electronic and or metallic implants in the skull or brain
9. Current medication use known to alter HD-tDCS reactivity

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Rey Auditory Verbal Learning Test Score | Baseline and immediately after completion of each HD-tDCS condition
  The RAVLT is a verbal episodic memory test that is sensitive to mesial and lateral verbal episodic memory circuit dysfunction. The primary outcome measure for this task is the total number of items immediately recalled during the learning trials and after the 20 minute delayed recall trial. Changes in scores from baseline to testing immediately following the completion of each condition will be examined.

SECONDARY OUTCOMES:
Changes in Delis Kaplan Executive Function System (DKEFS) Trail Making Test | Baseline and immediately after completion of each HD-tDCS condition
  The DKEFS Trail Making Test is a measure of cognitive flexibility and executive functions. The task requires the subject to as quickly as possible complete five conditions, involving number cancellation, number sequencing, letter sequencing, number-letter switching, and line tracing. The outcome measure for this task is the time to complete each of the five conditions. Changes in scores from baseline to testing immediately following the completion of each condition will be examined.
Changes in Delis Kaplan Executive Function System (DKEFS) Color-Word Interference Test | Baseline and immediately after completion of each HD-tDCS condition
  The DKEFS Color-Word Interference test is a measure of information processing speed and complex attention. The task requires the subject to as quickly as possible complete four conditions, involving color naming, word reading, response inhibition, and then switching back-and-forth between two response patterns. The outcome measure for this task is the time to complete each of the four conditions. Changes in scores from baseline to testing immediately following the completion of each condition will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States